CLINICAL TRIAL: NCT01342913
Title: A 12-week Study to Evaluate the 24 Hour Pulmonary Function of Fluticasone Furoate (FF)/Vilanterol Inhalation Powder (FF/VI Inhalation Powder) Once Daily Compared With Salmeterol/Fluticasone Propionate (FP) Inhalation Powder Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate the 24 Hour Spirometric Effect (FEV1) of Fluticasone Furoate/Vilanterol Inhalation Powder (100mcg Fluticasone Furoate (FF)/25mcg Vilanterol (VI)) Compared With Salmeterol/Fluticasone Propionate Inhalation Powder (50mcg Salmeterol/500mcg Fluticasone Propionate (FP))
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113107
Record Dates: First submitted 2011-04-14; First posted 2011-04-27 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/Vilanterol (Experimental): Inhaled Corticosteroid (ICS)/Long Acting Beta Agonist (LABA)
  Interventions: Drug: Fluticasone Furoate 100mcg/Vilanterol 25mcg
- Fluticasone Propionate/Salmeterol (Active Comparator): Inhaled Corticosteroid (ICS)/Long Acting Beta Agonist (LABA
  Interventions: Drug: Fluticaosne Propionate 500mcg/Salmeterol 50mcg

INTERVENTIONS:
Drug: Fluticasone Furoate 100mcg/Vilanterol 25mcg — Inhalation Powder
  Arms: Fluticasone Furoate/Vilanterol
Drug: Fluticaosne Propionate 500mcg/Salmeterol 50mcg — Inhalation Powder
  Arms: Fluticasone Propionate/Salmeterol

SUMMARY:
The purpose of this study is to evaluate the 24-hour spirometry effect (FEV1) of Fluticasone Furoate/Vilanterol 100/25mcg once daily compared with Salmeterol/Fluticasone Propionate 50/500mcg twice daily over a 12-week treatmen period in subjects with COPD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, multi-centre parallel group study. Subjects who meet the eligilibilty criteria at Screening and meet the randomization criteria at the end of a 2-week Run-In period will enter a 12-week Treatment period. There will be a 7-day Follow-up period after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Male or females ≥ 40 years of age
* Established clinical history of COPD by ATS/ERS definition
* Females are eligible to enter and participate if of non-childbearing potential, or if of child bearing potential, has a negative serum pregnancy test at screening, and agrees to one of the acceptable contraceptive methods listed in protocol, used consistently and correctly
* Former or current smoker > 10 pack years
* Post-albuterol spirometry criteria: FEV1/FVC ratio ≤ 0.70 and FEV1 ≤ 70% of predicted normal (NHANES III)
* have been hospitalised or have been treated with oral corticosteroids or antibiotics for their COPD within the last 3 years prior to Screening (Visit 1)

Exclusion Criteria:

* Current diagnosis of asthma
* Subjects with other respiratory disorders including active tuberculosis, α1-antitrypsin deficiency, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung volume reduction surgery within previous 12 months
* Clinically significant abnormalities not due to COPD by chest x-ray
* Hospitalized for poorly controlled COPD within 12 weeks of Screening
* Poorly controlled COPD 6 weeks prior to Screening, defined as acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician
* Lower respiratory infection requiring antibiotics 6 weeks prior to Screening
* Uncontrolled or clinically significant (in opinion of PI) cardiovascular, hypertension, neurological, psychiatric, renal, hepatic, immunological, endocrine, peptic ulcer disease, or hematological abnormalities
* Carcinoma not in complete remission for at least 5 years
* Subjects with history of hypersensitivity to study medications (e.g., beta-agonists, corticosteroid) or components of inhalation powder (e.g., lactose, magnesium stearate)
* Subjects with history of severe milk protein allergy that, in opinion of study physician, contraindicates subject's participation - Known/suspected history of alcohol or drug abuse in the last 2 years
* Women who are pregnant or lactating or plan to become pregnant
* Subjects medically unable to withhold albuterol and/or ipratropium 4 hours prior to spirometry testing at each study visit
* Use of certain medications such as bronchodilators and corticosteroids for the protocol-specific times prior to Visit 1 (the Investigator will discuss the specific medications)
* Long Term Oxygen Therapy (LTOT) or nocturnal oxygen therapy >12 hours a day
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening or during the study - Non-compliance or inability to comply with study procedures or scheduled visits
* Affiliation with investigator site

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2011-02-01; Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- Belgium (6):
  - GSK Investigational Site, Bouge
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Gilly
- France (7):
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Pessac
- Germany (9):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (9):
  - GSK Investigational Site, Acquaviva Delle Fonti BA, Apulia
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Sesto S. Giovanni MI, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Cittadella PD, Veneto
  - GSK Investigational Site, Verona, Veneto
- Philippines (3):
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Lipa City
  - GSK Investigational Site, Quezon City
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Piekary Śląskie
  - GSK Investigational Site, Wilkowice
- Russia (5):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Yaroslavl
- Spain (7):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Valencia
- Ukraine (5):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Agusti A, de Teresa L, De Backer W, Zvarich MT, Locantore N, Barnes N, Bourbeau J, Crim C. A comparison of the efficacy and safety of once-daily fluticasone furoate/vilanterol with twice-daily fluticasone propionate/salmeterol in moderate to very severe COPD. Eur Respir J. 2014 Mar;43(3):763-72. doi: 10.1183/09031936.00054213. Epub 2013 Oct 10. PMID 24114969
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1, participants entered a 2-week, single-blind (placebo) Run-in Period to obtain Baseline assessments of salbutamol use and to evaluate adherence with study treatment and procedures, diary card completion, and assessment of disease stability. At Visit 2, participants were randomized to a 12-week, double-blind Treatment Period.
Groups:
- Placebo + Salbutamol: Participants were instructed to take single-blind placebo (ACCUHALER/DISKUS and Novel Dry Powder Inhaler [NDPI]): one inhalation each morning from each device, and one inhalation from the ACCUHALER/DISKUS in the evening. In addition, all participants received supplemental albuterol (salbutamol) (metered dose inhaler [MDI] and/or nebules) to be used on an as-needed basis. Ipratropium bromide alone was permitted, provided that the participant was on a stable dose from Visit 1 (Screening) and remained on the stable dose throughout the study; however, ipratropium must have been withheld for 4 hours prior to and during each clinic visit.
- Salmeterol/FP 50/500 µg BID: Participants received a Salmeterol and Fluticasone Propionate (FP) 50/500 microgram (µg) inhalation (available as a combination dry inhalation powder of Salmeterol 50 µg and FP 500 µg in single strip) twice daily (BID) (morning and evening) from the ACCUHALER/DISKUS and placebo once daily (QD) in the morning from the NDPI over the course of 12 weeks.
- FF/VI 100/25 µg QD: Participants received a Fluticasone Furoate /Vilanterol (FF/VI) 100/25 µg inhalation (available as dry inhalation powder in two separate strips of FF 100 µg and VI 25 µg) QD in the morning from the NDPI and placebo BID (morning and evening) from the ACCUHALER/DISKUS over the course of 12 weeks.
Period: 2-week Run-in Period
Arm/Group | Placebo + Salbutamol | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Started | 702 | 0 | 0
Completed | 528 | 0 | 0
Not Completed | 174 | 0 | 0
Not completed — Inclusion/Exclusion Criteria Not Met | 66 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Continuation Criteria Not Met | 88 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Placebo + Salbutamol | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Started | 0 | 262 | 266
Completed | 0 | 246 | 243
Not Completed | 0 | 16 | 23
Not completed — Adverse Event | 0 | 3 | 6
Not completed — Lack of Efficacy | 0 | 2 | 3
Not completed — Protocol Violation | 0 | 6 | 9
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD | Total
Number analyzed (Participants) | 262 | 266 | 528
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.07) | 63.0 (8.10) | 62.9 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 54 | 95
  Male | 221 | 212 | 433
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 1 | 0 | 1
  Asian-South East Asian Heritage | 53 | 48 | 101
  White-Arabic/North African Hertage | 2 | 1 | 3
  White/Caucasian/European Heritage | 206 | 217 | 423

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Trough in 24-hour Weighted-mean FEV1 on Treatment Day 84
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1). The weighted mean was calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5, 15, 30, and 60 minutes (min) and 2, 4, 6, 8, 12, 13, 14, 16, 20, and 24 hours on Treatment Day 84. Baseline trough FEV1 was the mean of the two assessments made 30 and 5 minutes pre-dose on Treatment Day 1. Change from Baseline was calculated as the average of the Day 84 values minus the Baseline value.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least 1 dose of double-blind medication. Randomized participants were assumed to have received double-blind medication unless definitive evidence to the contrary existed. Only participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Number analyzed (Participants) | 233 | 224
Liters | 0.108 (0.0145) | 0.130 (0.0148)
Statistical Analysis 1: Comparison: Salmeterol/FP 50/500 µg BID vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.282, ANCOVA; Least squares mean difference = 0.022, 95% CI 2-sided [-0.018 to 0.063]

2. Secondary Outcome: Time to Onset on Treatment Day 1
Description: Time to onset on Treatment Day 1 is defined as the time to an increase of 100 milliliters (mL) from Baseline in FEV1. Time of onset was calculated over 0 to 4 hours (5 min, 15 min, 30 min, 60 min, 120 min, and 240 min) post-dose.
Time Frame: Day 1
Population: ITT Population. Only participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Number analyzed (Participants) | 260 | 260
Minutes | 28 [5 to 240] | 16 [5 to 240]

3. Secondary Outcome: Change From Baseline in Trough FEV1 on Treatment Day 85
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1). Trough FEV1 was defined as the 24-hour FEV1 assessment, which was obtained on Day 85. Baseline is defined as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1.Change from Baseline was calculated as the average of the Day 85 values minus the Baseline value.
Time Frame: Baseline and Day 85
Population: Only participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Number analyzed (Participants) | 245 | 242
Liters | 0.088 (0.0154) | 0.111 (0.0155)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 12 weeks).
Description: All AEs and SAEs were followed until resolution, until the condition stabilized, until the event was otherwise explained, or until the participant was lost to follow-up.
Arm/Group | Salmeterol/FP 50/500 µg BID | FF/VI 100/25 µg QD
Serious Adverse Events (participants affected / at risk) | 3/262 | 6/266
Other Adverse Events (participants affected / at risk) | 30/262 | 32/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol/FP 50/500 µg BID (N=262) | FF/VI 100/25 µg QD (N=266)
Pneumonia (Infections and infestations) | 2 | 1
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol/FP 50/500 µg BID (N=262) | FF/VI 100/25 µg QD (N=266)
Headache (Nervous system disorders) | 18 | 20
Nasopharyngitis (Infections and infestations) | 12 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.